CLINICAL TRIAL: NCT05448443
Title: Crossover, Double-blind, Phase 2 Study of AD981 Versus Placebo in Obesity Hypoventilation Syndrome
Brief Title: Study of AD981 Versus Placebo in Obesity Hypoventilation Syndrome
Acronym: ATOHS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Apnimed Inc. (Unknown); VIS Ethic Research Srl (Unknown); University of Florence (Other); STM Pharma PRO srl (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09J201
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Obesity Hypoventilation Syndrome (OHS)
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Intervention Model Description: Patients who meet the eligibility criteria will be randomized equally to receive AD981 or matching placebo.
  After 14 days of treatment and a washout period, the patients crossover to the other treatment arm for 14 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD981 (Experimental): AD981
  Interventions: Drug: AD981
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AD981 — Oral administration of AD981 in the morning and before sleep for 14 days
  Arms: AD981
Other: Placebo — Oral administration of placebo in the morning and before sleep for 14 days
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled, cross-over, phase II, single center efficacy study of AD981 in patients with obesity hypoventilation syndrome documented by polysomnography (PSG) and transcutaneous, overnight measurement of CO2 (PtcCO2).

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand the nature of the study and sign the informed consent
* BMI > 35 kg/m2 and presence of nocturnal hypoventilation
* Previous surgical treatment for OSA is allowed if ≥ 1 year prior to enrollment
* If in treatment, CPAP or BPAP or mandibular advancement device or positional therapy intolerance or poor compliance

Exclusion Criteria:

* Narcolepsy, craniofacial malformation, renal failure, hepatic disease, schizophrenia, schizoaffective disorder or bipolar disorder, cognitive dysfunction, severe neurological disorder, pheochromocytoma, adrenocortical insufficiency, hyperchloremic acidosis.
* Respiratory (COPD, ILD, oxygen therapy) or cardiac (Heart Failure, Atrial fibrillation, established severe peripheral arterial disease) disease or hypertension requiring more than 3 medications for control
* Cardiomyopathies, heart malformation or structural heart alterations, severe rhythm disorders, established coronary heart disease or other cardiac conditions, which could determine sudden death
* Attempted suicide or suicidal ideation
* Drugs of abuse or substance use disorder
* A significant illness or infection requiring medical treatment in the past 30 days.
* Untreated narrow angle glaucoma.
* Women who are pregnant or nursing.
* Treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors, or monoamine oxidase inhibitors (MAOI) or linezolid within 14 days of the start of treatment, allergies to sulfonamides.
* Diabetes with unstable glucose control in the past 15 days.
* > 500 mg/day of Aspirin
* Low sodium or potassium.
* Any condition that in the investigator's opinion would present an unreasonable risk to the participant.
* History of using oral or nasal devices (such as mandibular advancement devices) for the treatment of OSA may enroll as long as the devices are not used during participation in the study for at least 2 weeks prior to study begin.
* History of using devices to affect participant sleeping position for the treatment of OSA, e.g. to discourage supine sleeping position, may enroll as long as the devices are not used during participation in the study.
* Use of another investigational agent within 30 days or 5 half-lives, whichever is longer, prior to dosing.
* Patient currently receiving: MAOIs, Serotonin and Norepinephrine Reuptake Inhibitors, Norepinephrine Reuptake Inhibitors, Lithium, Tricyclic antidepressants, strong CYP2D6 inhibitors, other strong inhibitors cytochrome P450, thiazides diuretics, benzodiazepines, opioids, drugs with clinically significant cardiac QT-interval prolonging effects, drugs known to lower seizure threshold, amphetamines, antiepileptics, modafinil or armodafinil, beta2 agonists, antipsychotics, pseudoephedrine, phenylephrine, oxymetazoline, drugs for Parkinson's, Alzheimer's, Huntington's, Amyotrophic Lateral Sclerosis, or drugs for other neurodegenerative diseases, more than 500 mg/day of Aspirin or salicylates, sodium Phosphate.
* Known hypersensitivity to study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Nocturnal transcutaneous CO2 pressure (PtcCO2) | From baseline to the last day of treatment (14 days after the start of each treatment period)

SECONDARY OUTCOMES:
Proportion of participants without nocturnal hypoventilation | From baseline to the last day of treatment (14 days after the start of each treatment period)
Apnea-Hypopnea Index (AHI) | From baseline to the last day of treatment (14 days after the start of each treatment period)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Perger, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano,Ospedale San Luca, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perger E, Parati G, Faini A, Gell L, Faverio P, Luppi F, Bertoli S, Brunani A, Bigagli E, Lombardi C, Taranto-Montemurro L. Acetazolamide Plus Atomoxetine for Obesity Hypoventilation Syndrome Treatment. Chest. 2025 Sep 25:S0012-3692(25)05384-X. doi: 10.1016/j.chest.2025.09.019. Online ahead of print. PMID 41015199